CLINICAL TRIAL: NCT03562806
Title: MRI 3D UTE Hyper-Cones & ZTE for PET/MR Lung Attenuation Correction & for Lung Diagnostic Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Tested MR sequence was inferior in preliminary evaluation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-00899
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MR (single arm) (Experimental): PET and MR sequence acquisition on SIGNA PET/MR device
  Interventions: Diagnostic Test: PET/MR image acquisition

INTERVENTIONS:
Diagnostic Test: PET/MR image acquisition — Acquisition of PET and MR sequences on SIGNA PET/MR device.

SUMMARY:
MRI 3D UTE Hyper-Cones & ZTE for PET/MR lung attenuation correction & for lung diagnostic imaging

DETAILED DESCRIPTION:
The primary objective is to clinically test the feasibility of 3D UTE Hyper-Cones & ZTE in capturing lung density of patients with lung diseases at reasonable clinical imaging times compared to standard MR lung protocols (LAVA-Flex, PROPELLER). Secondly, we want to investigate if Hyper-Cones & ZTE can be used for lung imaging such as vessels and air-pathways, oncological patients, lung nodules and lung infiltration & parenchyma pathophysiology such as chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* informed consent and signature
* clinical PET/CT planned and performed at Wagi site in Schlieren
* male or female patients
* from 18 to 80 years of age.

Exclusion Criteria:

- same exclusion criteria as for the clinical PET/CT exam (i.e. pregnant women).

Additional exclusion criteria:

- standard exclusion criteria for clinical MRI (evaluated by clinical standard determined by MRI questionnaire).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Confirm that lung density map extraction is feasible through Hyper-Cones & ZTE scanning. | 1 year
  Confirm that lung density map extraction is feasible through Hyper-Cones & ZTE scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Huellner, M.D., Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Department of Nuclear Medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No